CLINICAL TRIAL: NCT06382480
Title: Meal Timing-based Strategies to Improve Glucose Metabolism in Prediabetes and Type 2 Diabetes
Brief Title: PROTeIn-rich Meals to Control Glucose
Acronym: PROTIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Charite University, Berlin, Germany (Other); Helmholtz Center Munich (Unknown); Hasso Plattner Institute, Potsdam, Germany (Unknown)
Responsible Party: Principal Investigator, Olga Ramich (formerly Pivovarova), Head of Research Group Molecular Nutritional Medicine, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 90/2023
Record Dates: First submitted 2024-03-15; First posted 2024-04-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Overweight; Obesity; Prediabetes; Type 2 Diabetes
Keywords: Glucose; Overweight; Obesity; Prediabetes; Type 2 Diabetes; Metabolism; Chrononutrition; Macronutrient composition; High-protein; High-carb; Isocaloric diet; Prevention and treatment of type 2 diabetes
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Intervention Model Description: The trial will have a cross-over design and compare metabolic effects of two isocaloric 4-week interventions with opposite timely distribution of macronutrient intake divided by a 4-week wash-out phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HP/HC - HC/HP (Experimental): Isocaloric 4-week HP/HC intervention followed by a 4-week HC/HP intervention.
  Interventions: Other: Diet with specific macronutrient composition.
- HC/HP - HP/HC (Experimental): Isocaloric 4-week HC/HP intervention followed by a 4-week HP/HC intervention.
  Interventions: Other: Diet with specific macronutrient composition.

INTERVENTIONS:
Other: Diet with specific macronutrient composition. — The intervention is about an isocaloric diet that differs in terms of distribution of carbohydrates and protein throughout the day. The interventions include a HP-breakfast and a HC-dinner vs. a HC-breakfast and a HP-dinner. A HP low-carb meal (breakfast or dinner) will contain 35%E protein, 35%E carbs, and 30%E fat, and a HC meal (breakfast or dinner) will contain 10%E protein, 60%E carbs, and 30%E fat.

SUMMARY:
The overall aim is to identify the dietary pattern for prevention and treatment of type 2 diabetes. The specific aim of this pilot project is to compare effects of two diets with different diurnal distribution of carbohydrates and protein on the glucose metabolism in subjects with prediabetes and type 2 diabetes and its effects on inflammatory status.

DETAILED DESCRIPTION:
Overweight individual with prediabetes and non-insulin treated type 2 diabetes will be recruited for the study. The trial will have a cross-over design and compare metabolic effects of two isocaloric 4-week interventions with opposite timely distribution of macronutrient intake - a high-protein (HP) breakfast and a high-carb (HC) dinner (HP/HC intervention) vs. a HC breakfast and a HP dinner (HC/HP intervention) - divided by a 4-week wash-out phase. A HP low-carb meal (breakfast or dinner) will contain 35%E protein, 35%E carbs, and 30%E fat, and a HC meal (breakfast or dinner) will contain 10E%protein, 60%E carbs, and 30%E fat.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes (fasting blood sugar 100-125 mg/dl)
* Diabetes type 2 (fasting blood sugar >126 mg/dl)
* Overweight and obesity (BMI 25-50 kg/m2)

Exclusion Criteria:

* Other diabetes types
* Insulin treatment
* Shift work
* Weight changes >5% within past 3 months
* Systemic glucocorticoid therapy
* Systemic infections
* Severe anemia
* High blood pressure (>180/110 mmHg)
* Endocrinologic, liver and heart disorders
* Immune diseases
* Thyroid dysfunction
* Heart attack or stroke
* Cancer in the last 2 years
* Eating disorders, food intolerance/allergy, addiction disorders, digestive disorders intestinal, liver, cardiovascular diseases
* Hereditary or acquired coagulation disorders
* Non-interruptible intake of blood thinners (anticoagulants)
* Specific diets, intermittent fasting
* Pregnancy or breastfeeding
* Severe internal or psychiatric disorders or other conditions and drugs therapy that might influence the outcome of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour glucose | 4 weeks
  Mean 24-hour glucose assessed by continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Measurement of height | 4 weeks
  Height measured by stadiometer
Measurement of body weight | 4 weeks
  Body weight measured by body scale
Waist and hip circumference / waist to hip ratio | 4 weeks
  Waist and hip circumference measured by tape measure
Systolic and diastolic blood pressure | 4 weeks
  Systolic and diastolic blood pressure changes measurement by manometer
Body fat and lean mass | 4 weeks
  Body fat and lean mass assessed by bioelectrical impendance analysis (BIA)
Energy expenditure and substrate oxidation rates | 4 weeks
  Energy expenditure and substrate oxidation rates assessed by indirect calorimetry
Hepatic values (gamma-glutamyl transferase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT)) | 4 weeks
  GGT, AST, ALT etermined in fasting blood samples
Renal values (creatinine, urea, uric acid) | 4 weeks
  Renal values determined in fasting blood samples
Intra- und inter-day glycemic variability | 4 weeks
  Indices of intra- and inter-day glycemic variability assessed by continuous glucose monitoring (CGM)
Glucose levels in meal tolerance test (MTT) | 4 weeks
  Glucose levels in blood samples collected in MTT
Metabolic hormones (insulin, C-peptide, glucagon, glucagon-like peptite 1(GLP-1), gastric inhibitory polypeptide (GIP), peptide YY (PYY), ghrelin, adiponectin, leptin) | 4 weeks
  Blood levels of metabolic hormones assessed in fasting state and during the MTT
Inflammatory markers and T cell populations analyses | 4 weeks
  Level of the inflammatory markers IL-6, TNFa, MCP-1 and T cell populations in circulation and adipose tissue are assessed through blood analysis and fat biopsy
Satiety and hunger scores | 4 weeks
  Satiety and hunger scores assessed using Visual Analog Scale (VAS with a scale of 1-100, where higher values correspond to stronger satiety/hunger)
Sleep/wake timing and sleep quality | 4 weeks
  Sleep/wake timing and sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI score, which ranges from 0-21, where higher values correspond to worse sleep quality) and also monitored by an ActiGraph device
Physical activity | 4 weeks
  24-h physical activity will be monitored by an ActiGraph device
Adipose tissue transcriptome | 4 weeks
  RNA-Seq analysis of subcutaneous adipose tissue sample
Gene expression in peripheral blood mononuclear cells (PBMC) | 4 weeks
  Expression of metabolic genes assessed by qPCR
Gut microbiota and microbiome-derived metabolites | 4 weeks
  Determined in stool samples and blood plasma
Determination of decision behavior | 4 weeks
  Impulsiveness assessed by decision making tasks on computer

CONTACTS AND LOCATIONS:
Overall Officials: Olga Ramich, PD Dr., Principal Investigator — German Institute of Human Nutrition
Locations (1):
- Olga Ramich, Potsdam, Potsdam-Rehbrücke, Germany

IPD SHARING:
Plan to Share IPD: No